CLINICAL TRIAL: NCT05258318
Title: Double Rewire Versus Double Kissing Crush Stenting Technique in Left Main Bifurcation Lesions
Acronym: DR vs DK crush
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Low recruitment rate
Sponsor: Fundación EPIC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EPIC20-DR vs DK crush
Record Dates: First submitted 2022-02-17; First posted 2022-02-28 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2022-02

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DR crush technique (Active Comparator)
  Interventions: Procedure: DR crush
- DK crush technique (Experimental)
  Interventions: Procedure: DK crush

INTERVENTIONS:
Procedure: DK crush — Double Kissing Crush (DK-Crush) technique in patients with Unprotected Left Main Bifurcation lesions (ULMb).
  Arms: DK crush technique
Procedure: DR crush — Double Rewire crush technique (DR-Crush) in patients with Unprotected Left Main Bifurcation lesions (ULMb).
  Arms: DR crush technique

SUMMARY:
The DR vs DK trial is designed to elucidate the benefits of Double Rewire crush technique (DR-Crush) over Double Kissing Crush (DK-Crush) technique in patients with Unprotected Left Main Bifurcation lesions (ULMb).

DETAILED DESCRIPTION:
DR vs DK is a multicentre, randomized, prospective, non-inferiority clinical trial designed to evaluate the efficacy and safety of DR crush over DK crush for patients with ULMb. More than 12 tertiary centres from Spain will participate including patients. Subjects with Medina 1,1,1 ULMb will be randomized in a 1:1 fashion to DR or DK crush. In order to avoid bias, the Sirolimus coronary stent will be used in all patients (UltimasterTM TanseiTM). The use of Intracoronary imaging techniques are recommended. The primary endpoint is target lesion failure (TLF) including target vessel myocardial infarction, cardiac death and TLR. Other endpoints address individual event of primary end-point, and target vessel revascularization. The safety objective is the ST. Recruitment began in January 2022 and will be completed in January 2024; 180 patients will be randomized.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18-90 years of age.
* Patients who gave written informed consent for participation in the trial.
* Lesions are eligible for percutaneous coronary intervention (PCI).
* Patient has stable/unstable angina or myocardial infarction (MI): all-comers.
* ULMb (Medina 1,1,1) with/without left main ostial/shaft lesions. Downstream lesions in LAD or LCX could be covered by two stents. Severe calcification needing rotational atherectomy, orbital atherectomy or Laser are included.
* Diameter stenosis in LAD/LM and LCX ≥ 50% by visual estimation or minimal luminal area by IVUS in LM ≤6 mm2.

Exclusion Criteria:

* Restenotic lesions.
* Patient was allergic to the study stent or protocol-required concomitant medications.
* Patient is intolerable to dual anti-platelet therapy.
* Patient has any other serious medical illness that may reduce life expectancy to <12 months.
* Patient is a woman who is pregnant or nursing.
* Patient has a planned procedure that may cause non-compliance with the protocol or confound data interpretation.
* Patient is participating in another clinical trial.
* Patients in shock.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-02-20 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Rate of target vessel failure | 12 months
  as the composite of cardiac death, target vessel myocardial infarction (TVMI), and clinically driven TVR.
Rate of stent thrombosis | 12 months
  The safety endpoint was stent thrombosis (ST), according to the definition by Academic Research Consortium.

SECONDARY OUTCOMES:
Rate of MACE | 1 month
  as the composite of cardiac death, non-fatal target vessel myocardial infarction (TVMI), and unplaned target vessel revascularization
Rate of MACE | 12 months
  as the composite of cardiac death, non-fatal target vessel myocardial infarction (TVMI), and unplaned target vessel revascularization

REFERENCES:
- [Background] Steigen TK, Maeng M, Wiseth R, Erglis A, Kumsars I, Narbute I, Gunnes P, Mannsverk J, Meyerdierks O, Rotevatn S, Niemela M, Kervinen K, Jensen JS, Galloe A, Nikus K, Vikman S, Ravkilde J, James S, Aaroe J, Ylitalo A, Helqvist S, Sjogren I, Thayssen P, Virtanen K, Puhakka M, Airaksinen J, Lassen JF, Thuesen L; Nordic PCI Study Group. Randomized study on simple versus complex stenting of coronary artery bifurcation lesions: the Nordic bifurcation study. Circulation. 2006 Oct 31;114(18):1955-61. doi: 10.1161/CIRCULATIONAHA.106.664920. Epub 2006 Oct 23. PMID 17060387
- [Background] Latib A, Colombo A. Bifurcation disease: what do we know, what should we do? JACC Cardiovasc Interv. 2008 Jun;1(3):218-26. doi: 10.1016/j.jcin.2007.12.008. PMID 19463303
- [Background] Ragosta M, Dee S, Sarembock IJ, Lipson LC, Gimple LW, Powers ER. Prevalence of unfavorable angiographic characteristics for percutaneous intervention in patients with unprotected left main coronary artery disease. Catheter Cardiovasc Interv. 2006 Sep;68(3):357-62. doi: 10.1002/ccd.20709. PMID 16892431
- [Background] Naganuma T, Chieffo A, Meliga E, Capodanno D, Park SJ, Onuma Y, Valgimigli M, Jegere S, Makkar RR, Palacios IF, Costopoulos C, Kim YH, Buszman PP, Chakravarty T, Sheiban I, Mehran R, Naber C, Margey R, Agnihotri A, Marra S, Capranzano P, Leon MB, Moses JW, Fajadet J, Lefevre T, Morice MC, Erglis A, Tamburino C, Alfieri O, Serruys PW, Colombo A. Long-term clinical outcomes after percutaneous coronary intervention versus coronary artery bypass grafting for ostial/midshaft lesions in unprotected left main coronary artery from the DELTA registry: a multicenter registry evaluating percutaneous coronary intervention versus coronary artery bypass grafting for left main treatment. JACC Cardiovasc Interv. 2014 Apr;7(4):354-61. doi: 10.1016/j.jcin.2013.11.014. Epub 2014 Mar 14. PMID 24630886
- [Background] Carrie D, Eltchaninoff H, Lefevre T, Silvestri M, Levy G, Maupas E, Brunel P, Fajadet J, Le Breton H, Gilard M, Blanchard D, Glatt B; FRIEND. Twelve month clinical and angiographic outcome after stenting of unprotected left main coronary artery stenosis with paclitaxel-eluting stents--results of the multicentre FRIEND registry. EuroIntervention. 2009 Jan;4(4):449-56. doi: 10.4244/eijv4i4a78. PMID 19284066
- [Background] Ali WE, Vaidya SR, Ejeh SU, Okoroafor KU. Meta-analysis study comparing percutaneous coronary intervention/drug eluting stent versus coronary artery bypass surgery of unprotected left main coronary artery disease: Clinical outcomes during short-term versus long-term (> 1 year) follow-up. Medicine (Baltimore). 2018 Feb;97(7):e9909. doi: 10.1097/MD.0000000000009909. PMID 29443766
- [Background] Stone GW, Sabik JF, Serruys PW, Simonton CA, Genereux P, Puskas J, Kandzari DE, Morice MC, Lembo N, Brown WM 3rd, Taggart DP, Banning A, Merkely B, Horkay F, Boonstra PW, van Boven AJ, Ungi I, Bogats G, Mansour S, Noiseux N, Sabate M, Pomar J, Hickey M, Gershlick A, Buszman P, Bochenek A, Schampaert E, Page P, Dressler O, Kosmidou I, Mehran R, Pocock SJ, Kappetein AP; EXCEL Trial Investigators. Everolimus-Eluting Stents or Bypass Surgery for Left Main Coronary Artery Disease. N Engl J Med. 2016 Dec 8;375(23):2223-2235. doi: 10.1056/NEJMoa1610227. Epub 2016 Oct 31. PMID 27797291
- [Background] Holm NR, Makikallio T, Lindsay MM, Spence MS, Erglis A, Menown IBA, Trovik T, Kellerth T, Kalinauskas G, Mogensen LJH, Nielsen PH, Niemela M, Lassen JF, Oldroyd K, Berg G, Stradins P, Walsh SJ, Graham ANJ, Endresen PC, Frobert O, Trivedi U, Anttila V, Hildick-Smith D, Thuesen L, Christiansen EH; NOBLE investigators. Percutaneous coronary angioplasty versus coronary artery bypass grafting in the treatment of unprotected left main stenosis: updated 5-year outcomes from the randomised, non-inferiority NOBLE trial. Lancet. 2020 Jan 18;395(10219):191-199. doi: 10.1016/S0140-6736(19)32972-1. Epub 2019 Dec 23. PMID 31879028
- [Background] Morice MC, Serruys PW, Kappetein AP, Feldman TE, Stahle E, Colombo A, Mack MJ, Holmes DR, Choi JW, Ruzyllo W, Religa G, Huang J, Roy K, Dawkins KD, Mohr F. Five-year outcomes in patients with left main disease treated with either percutaneous coronary intervention or coronary artery bypass grafting in the synergy between percutaneous coronary intervention with taxus and cardiac surgery trial. Circulation. 2014 Jun 10;129(23):2388-94. doi: 10.1161/CIRCULATIONAHA.113.006689. Epub 2014 Apr 3. PMID 24700706
- [Background] Zhang D, He Y, Yan R, Yin D, Feng L, Xu B, Yang Y, Zhu C, Dou K. A novel technique for coronary bifurcation intervention: Double rewire crush technique and its clinical outcomes after 2 years of follow-up. Catheter Cardiovasc Interv. 2019 Feb 15;93(S1):851-858. doi: 10.1002/ccd.28066. Epub 2019 Jan 2. PMID 30604485
- [Background] Chen SL, Xu B, Han YL, Sheiban I, Zhang JJ, Ye F, Kwan TW, Paiboon C, Zhou YJ, Lv SZ, Dangas GD, Xu YW, Wen SY, Hong L, Zhang RY, Wang HC, Jiang TM, Wang Y, Chen F, Yuan ZY, Li WM, Leon MB. Comparison of double kissing crush versus Culotte stenting for unprotected distal left main bifurcation lesions: results from a multicenter, randomized, prospective DKCRUSH-III study. J Am Coll Cardiol. 2013 Apr 9;61(14):1482-8. doi: 10.1016/j.jacc.2013.01.023. Epub 2013 Mar 10. PMID 23490040
- [Background] Chen SL, Zhang JJ, Han Y, Kan J, Chen L, Qiu C, Jiang T, Tao L, Zeng H, Li L, Xia Y, Gao C, Santoso T, Paiboon C, Wang Y, Kwan TW, Ye F, Tian N, Liu Z, Lin S, Lu C, Wen S, Hong L, Zhang Q, Sheiban I, Xu Y, Wang L, Rab TS, Li Z, Cheng G, Cui L, Leon MB, Stone GW. Double Kissing Crush Versus Provisional Stenting for Left Main Distal Bifurcation Lesions: DKCRUSH-V Randomized Trial. J Am Coll Cardiol. 2017 Nov 28;70(21):2605-2617. doi: 10.1016/j.jacc.2017.09.1066. Epub 2017 Oct 30. PMID 29096915
- [Background] Chen SL, Santoso T, Zhang JJ, Ye F, Xu YW, Fu Q, Kan J, Paiboon C, Zhou Y, Ding SQ, Kwan TW. A randomized clinical study comparing double kissing crush with provisional stenting for treatment of coronary bifurcation lesions: results from the DKCRUSH-II (Double Kissing Crush versus Provisional Stenting Technique for Treatment of Coronary Bifurcation Lesions) trial. J Am Coll Cardiol. 2011 Feb 22;57(8):914-20. doi: 10.1016/j.jacc.2010.10.023. PMID 21329837
- [Background] Chen SL, Ye F, Zhang JJ, Xu T, Tian NL, Liu ZZ, Lin S, Shan SJ, Ge Z, You W, Liu YQ, Qian XS, Li F, Yang S, Kwan TW, Xu B, Stone GW. Randomized Comparison of FFR-Guided and Angiography-Guided Provisional Stenting of True Coronary Bifurcation Lesions: The DKCRUSH-VI Trial (Double Kissing Crush Versus Provisional Stenting Technique for Treatment of Coronary Bifurcation Lesions VI). JACC Cardiovasc Interv. 2015 Apr 20;8(4):536-46. doi: 10.1016/j.jcin.2014.12.221. Epub 2015 Mar 26. PMID 25819187